CLINICAL TRIAL: NCT02282631
Title: The RIGHT TRACKS Study - Development and Feasibility of an Incentive Scheme to Promote Active School Travel in Year 5 Children
Brief Title: Development and Feasibility of an Incentive Scheme to Promote Walking/Cycling to School
Acronym: RIGHT_TRACKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Principal Investigator, Samuel Ginja, Mr Samuel Ginja, Newcastle University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AST-00759
Record Dates: First submitted 2014-09-05; First posted 2014-11-04 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Physical Activity
Keywords: active school travel; active travel; incentive scheme; children; school; behaviour change
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group school (Experimental): School where the incentive scheme will be run.
  Interventions: Behavioral: Incentive scheme
- Control group school (No Intervention): School with no intervention; ongoing advice on active school travel.

INTERVENTIONS:
Behavioral: Incentive scheme — Children who actively travel to school, full or partway, enter a weekly £5 voucher draw, whereby chances of winning are proportional to the number of trips as reported by the parent.
  Other Names: Incentive-scheme, lottery-based scheme, intervention
  Arms: Intervention group school

SUMMARY:
The aim of this study is to investigate whether an incentive scheme is a feasible approach to increase walking/cycling to school.

DETAILED DESCRIPTION:
This will be a feasibility study using a two-arm cluster randomised controlled design; the Year 5 group (and respective school) will be the unit of randomisation. Participants will be Year 5 pupils, aged 9-10.

Data will be collected throughout approximately three months. In total, assessments will be carried out over a nine week period, which excludes an interval week between baseline and the first intervention week, and half-term (school holidays).

All children in Year 5's in the selected schools will be approached to participate and will be allocated randomly (according to the school they attend) to the two arms: (i) intervention group taking part in the incentive scheme and (ii) control group receiving ongoing curricular advice on active travel.

Parents' participation consists in completing a socio-demographic questionnaire and consent form, and in completing a daily form (or answering daily text messages) reporting whether child has actively traveled to school (AST report) .

A number of schools will be invited to participate by email. A reply by post, phone or email to the lead researcher will be requested within two weeks, at the end of which pending schools will be contacted by phone to confirm their decision. Of those interested, two schools will be selected, ideally matched for characteristics such as location, free school meals and AST rates.

Once the two participating schools have been identified, a meeting in person will be arranged with each head teacher at a time/place of their choice.

The researcher will then visit the schools and introduce the RIGHT TRACKS study to the Year 5 class. After the study has been presented and questions answered, an information pack will be sent home in the pupil's school folder. This pack will include an information leaflet for child, an information leaflet for the parent/carer, a parent questionnaire, a participant information sheet and a consent form. Two of the points stressed are confidentiality and the freedom to drop out of the study at any time without giving justification. After reading and having the chance of asking questions (by phone/email to the lead researcher), parents will be required to formally consent (opt in procedure) to their and to their child's participation.

Parental questionnaires and consent forms are expected to be filled in at home but phone or email inquiries may be made to the researcher during working hours. Within one week after delivery, parents will be requested to return completed and signed documents to the researcher. Specific methods of distribution and collection will be decided with the school beforehand to accommodate local circumstances and preferences.

Questionnaire completion will be requested of parents, however only return of the signed consent form will be essential to determine the child's participation. In addition, participating children will complete an assent form in the classroom.

Baseline assessment Following the identification of participants, children in both schools will be given and instructed to wear an accelerometer on a waist band above the lateral hip over the ensuing seven days, from the moment they get up until they go to bed, except for water-based activities and certain sports.

Together with the accelerometer, the child will be given the parent AST report form, which he/she must take home and return at the end of the seven day period, completed by the parent, together with the accelerometer. Four questions will be asked to parents in the parent AST report form, in relation to each day of the week: e.g. "On Monday did your child walk or cycle to school, all or part of the journey?", "At what time did your child leave home?", "At what time did your child arrive at school?", "Did your child stop anywhere on the way? If yes, how long was the stop for? ____ minutes".

Upon collection of the accelerometer and completed parents AST report forms, children's AST form will be filled out in the classroom retrospectively in relation to the five previous school days (mornings). The only question to be asked to children in relation to the five days is: e.g. "On Monday did you walk or cycle to school, all or part of the journey?" At the end of the baseline week, those complying with the study protocol will be rewarded, as stated in advance on the information materials: a prompt return of the completed parent AST report form and undamaged accelerometer, and completed child AST report form in the classroom, will be essential requisites for receiving a £5 thank you voucher.

Intervention phase The next stage of the RIGHT TRACKS consists in testing the feasibility of the incentive scheme. Similar to baseline, the quality of data from the three sources - accelerometry, parental AST report and child self-report of AST - will be examined. In particular, the validity of parental and child-reported AST will be assessed vis-à-vis accelerometry, currently considered to be one of the gold-standards. However, parental report of AST will be used as the basis of the incentive scheme. Once again, in both intervention and control conditions, there will be a £5 thanks voucher for every child taking part in the measurement procedures, in compliance with the protocol. At the end of the study, a debrief sheet will be handed to all participants, including parents and children, and to the two head teachers.

Intervention group - incentive scheme The incentive scheme will be explained to the intervention group in an introductory session. Partway active trips will be given particular emphasis. Each subsequent session is anticipated to take no more than 25 minutes per week of the classroom time.

The incentive scheme run in the intervention school consists of a prize draw taking place once a week. The prize is a £5 shopping gift voucher valid in a number of high street shops. Chances of winning depend entirely on the number of "points": the number of active trips to school reported exclusively by the parent on the AST report form, through the same questions used at baseline. For each week day that they travel to school the child gets one point. This point is the equivalent to a ticket with the child's ID number that will then be entering the draw. Each child can earn between zero and five tickets per week, depending on the number of active travel trips to school reported by the parent. Discrepant numbers between parental reports and those reported by the child or recorded on the accelerometer are of great interest for measurement, but will be disregarded for the purposes of the draw. In the absence of the parent AST report, the child report may be use for point count, but the child will be reminded that the parental report will be necessary for the next draw.

A difference between baseline and intervention phase concerns the format of the parent AST report form, which may now be completed in writing as before, or by SMS text messages on the weeks the child is not wearing the accelerometer. Preference for either of the options can be stated in advance in the consent form. Parents will be asked to keep them, fill in and return on time every week (personally or via the child), as the programme proceeds. Mobile phone respondents will be notified daily by SMS, to which they can reply directly. Questions asked will be the same in the paper version and mobile phone. However, on the two weeks the child wears the accelerometer, all participants will be asked to use the parent AST report. When the child is not wearing the accelerometer, the only question asked on the parental form or text messages is whether the child walked/cycled to school all or part of the journey. For those wearing the accelerometer in the intervention school, the point will be credited as long as the first question is answered (i.e. if parent indicated whether child actively traveled but failed to complete questions on times).

During the intervention phase, three tasks will be expected from children: (1) wearing an accelerometer for another seven-day period, which they must return to the classroom, together with the parent AST report form, (2) returning the parent AST report form in the remaining weeks (if applicable) and (3) complete an AST report form in the classroom each day of the draw.

Thank you vouchers (£5) will be issued on timely receipt of the accelerometer (together with AST forms), even if the accelerometer turns out to not have been worn for the requested time (i.e. at least four days, including at least one weekend day, and 10 hours each day).

The researcher will retire to a different room (or section of the school) and based on the parent AST report form only, points relative to the five previous days will be calculated. In the case of SMS, responses will be gathered in the evening, at the researcher's workplace, and next day's point will only be credited if received before 12noon (this will be stated in every text message that parents receive on a draw day). Class scores will be anonymously displayed on a graphic/chart week-after-week, in a printed version if possible or by hand if necessary. Depending on the school's preferences and availability, the logistics of counting points and producing tickets may be slightly different. For example, a teacher may agree to return all the completed parent AST reports to the school office in the morning, in which case the researcher could collect them and prepare the tickets in advance.

After producing all the tickets, the researcher will return to the classroom to distribute the accelerometers to the next batch of users. Once the thank you vouchers and accelerometers have been sorted out, the draw will finally take place in the classroom. A ticket will be picked out of a black string bag, probably by a school staff member of by the researcher. Depending on parental choice specified on the consent form, the incentive scheme voucher will be provided to the winner straight away, or will be left in the school office for later collection by the parent. The class score graphic/chart will be put on display on the wall.

Control group - normal curricular AST advice With the exception of the incentive scheme, identical procedures will be followed in both intervention and control groups. Each week, new groups of participants (e.g. the next five on the list) will be requested to wear the accelerometer, return the parent AST report form (if applicable) and complete their own AST report form.

Qualitative study One component of this study consists of semi-structured interviews with children, parents/carers and stakeholders, both from experimental and control groups, to explore different perspectives associated with the proposed intervention and trial procedures and to help refine both. Willingness to be interviewed will be expressed in the consent form before baseline in the case of parents (in addition to assent form in the case of children), from which a purposive sample will be selected based on the socio-demographic variables assessed in the questionnaire. The researcher will directly invite teachers and head teachers, who in turn will suggest other stakeholders for interview among their acquaintances (snowball sampling).

The aim will be to interview dropout participants throughout the intervention phase (as soon as they leave the study), and full participants immediately after the study has ended (January 2015). Sessions are expected to last between 30-45 minutes for adults and 15-30 minutes for children. Verbal consent to take part and to have the session audio-taped will be requested at the onset (in the case of children, to parents first and then by verbal assent), and the confidential nature of all records will be reiterated. Data will be securely stored in compliance with Newcastle University's regulations.

ELIGIBILITY:
Inclusion Criteria:

* Year 5 children in any of the selected schools
* Consent from parent and assent from child

Exclusion Criteria:

* No consent/assent

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine McColl, PhD, Study Director — Newcastle University; Bronia Arnott, PhD, Study Director — Newcastle University; Vera Araujo-Soares, PhD, Study Director — Newcastle University; Anil Namdeo, PhD, Study Director — Newcastle University; Samuel Ginja, MSc, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Institute of Health and Society, Baddiley-Clark Building, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ginja S, Arnott B, Araujo-Soares V, Namdeo A, McColl E. Feasibility of an incentive scheme to promote active travel to school: a pilot cluster randomised trial. Pilot Feasibility Stud. 2017 Nov 14;3:57. doi: 10.1186/s40814-017-0197-9. eCollection 2017. PMID 29167744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: School recruitment took place from late May 2014 to early July 2014. I emailed and phoned schools from my office, and then met personally with the two selected schools in mid July 2014.
  Family recruitment took place in mid September 2014. Invitations were distributed to children at school and returned by parents by post.
Pre-assignment Details: Recruitment of schools: one invitation email, second email two weeks later (reminder) and phone call (one week after reminder). Four schools replied positively out of 123 contacted (3.3%).
  Recruitment of participants: 29 (33.0%) returned a valid consent form before baseline; 2 returned a consent form after the start of baseline and were excluded
Groups:
- Control Group School: School with no intervention (incentive scheme)
- Intervention Group School: School with intervention (incentive scheme)
Period: Overall Study
Arm/Group | Control Group School | Intervention Group School
Started | 14 (The two dropouts happened on the 2nd and 3rd weeks post-baseline, respectively) | 15
Completed | 12 | 15
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control School: School with no intervention; ongoing advice on active school travel.
- Intervention School: School where the incentive scheme will be run.
  Incentive scheme: Children who actively travel to school, full or partway, enter a weekly £5 voucher draw. Every trip to school reported by the parent as being active (walking/cycling) corresponds to one ticket entered into the draw. In total, one child can have up to five tickets entered into one draw.
- Total: Total of all reporting groups
Arm/Group | Control School | Intervention School | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years of age] | 9 [9 to 9] | 9 [9 to 9] | 9 [9 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 5 | 8 | 13
Ethnic group [Number; unit: participants]
  White British | 13 | 14 | 27
  Other Ethnic Group | 1 | 1 | 2
Car available to drive child to school [Count of Participants; unit: Participants] | 9 | 12 | 21
Parent completing questionnaire has degree or higher degree [Count of Participants; unit: Participants] | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Schools Who Accepted to Take Part
Description: Percentage of schools who accepted to take part in this study
Time Frame: May 2014 to June 2014
Population: 123 schools were approached; 4 accepted to take part but only 2 were selected to take part
Measure: Number; unit: % schools who accepted to take part
Groups:
- Schools Contacted: Primary schools (or equivalent) located in the North East approached in this study
Arm/Group | Schools Contacted
Number analyzed (Participants) | 123
% schools who accepted to take part | 3.3

2. Primary Outcome: School Retention
Description: % of schools who were retained for the whole duration of the study (out of the two who took part)
Time Frame: September 2014 to December 2014
Measure: Number; unit: % schools retained for the whole study
Groups:
- Schools Who Took Part: Schools who took part in this study (two)
Arm/Group | Schools Who Took Part
Number analyzed (Participants) | 2
% schools retained for the whole study | 100

3. Primary Outcome: Recruitment of Participants
Description: Number of participants recruited in this study.
Time Frame: Sep 2014 to December 2014
Population: Number of participants approached to take part in the study
Measure: Number; unit: N of children who took part in the study
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 48 | 40
N of children who took part in the study | 14 | 15

4. Primary Outcome: Retention of Participants
Description: Number of participants who remained in the study until the end.
Time Frame: September 2014 to December 2014
Population: There were 14 participants in the control school, and 15 participants in the intervention school, at baseline. In the post-baseline weeks, there were two dropouts in the control school, and none in the intervention school.
Measure: Number; unit: N children retained for the whole study
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
N children retained for the whole study | 12 | 15

5. Primary Outcome: Number of Participants Who Returned Their Accelerometers on Time at the End of the Baseline Week
Description: Number of participants who returned their accelerometer to the researcher on the designated day, at end of baseline week (all children wore the accelerometer at the same time)
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Participants | 11 | 15

6. Primary Outcome: Number of Participants Who Returned Their Accelerometers on Time at the End of the Post-baseline Week
Description: Number of participants who returned their accelerometer on time to the researcher (myself) on the designated day, at end of post-baseline week. This was the second week of wear for participants. Whereas all participants were assessed concurrently at baseline, different subsamples were assessed every week at post-baseline.
Time Frame: 8 weeks after baseline
Population: Participants who stayed long enough in the study to wear the accelerometer a second time, at post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 12 | 15
Participants | 8 | 12

7. Primary Outcome: Accelerometers Lost or Damaged
Description: Number of accelerometers lost or damaged in this study
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Measure: Number; unit: N of accelerometers lost or damaged
Units Other Than Participants: Total N times accelerometer was worn
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (Total N times accelerometer was worn) | 26 | 30
N of accelerometers lost or damaged | 0 | 0

8. Primary Outcome: Parental ATS Paper Reports Returned
Description: N parental ATS* paper reports returned to researcher(me)
  *Active Travel to School
  * Paper reports with at least 1 box had been ticked out of the five boxes on the form (there was 1 box for each day of the week).
  * ATS reports were collected weekly, i.e. on the baseline week and on each of the eight post-baseline weeks. Accelerometers were only used twice; once at baseline (1week) and once at post-baseline (1week).
  * Parental paper ATS reports were preferred by 6 families, but on the 2 accelerometer weeks all participants had to use a paper reports including usual SMS respondents. In contr. group: all used paper reports at baseline (1st accel. week) (n=14), 6 usual paper respondents at post-baseline (6x8 weeks = 48), 6 SMS respondents who had to paper-report on the 2nd accel.week (both dropouts were SMS respondents & left too early for a 2nd accel.), so total N possible paper reports 14 + 48 + 6=68. Int. school: 15 participants & 8 usual paper respondents, total=15 + (8 x 8) + 7=86
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: The above number of participants corresponds to all participants in each group. The overall N of units analysed takes into account that although only some participants (6 in CG; 8 in IG) had chosen to report ATS by paper reports at baseline, everybody was expected to report by ATS paper report on the two weeks where the accelerometer was worn.
Measure: Number; unit: N of parental ATS paper reports returned
Units Other Than Participants: N of parental ATS paper reports
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N of parental ATS paper reports) | 68 | 86
N of parental ATS paper reports returned | 36 | 78

9. Primary Outcome: Child ATS Reports Returned
Description: Number of child ATS* reports returned to the researcher (myself) throughout the study. Child ATS reports were always on paper.
  *Active Travel to School
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: N of child ATS reports (always on paper) - is the total number of child ATS reports that could have been returned to the researcher throughout the study
Measure: Number; unit: N child ATS reports returned
Units Other Than Participants: N of child ATS reports
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N of child ATS reports) | 112 | 135
N child ATS reports returned | 108 | 134

10. Primary Outcome: Agreement Between Parent and Child Reports
Description: Inter-rater agreement between parent and child ATS* reports
  *Active Travel to School
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Measure: Number (95% Confidence Interval); unit: Kappa score
Units Other Than Participants: N trips to school with both reports
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N trips to school with both reports) | 356 | 582
Kappa score | 0.264 [0.138 to 0.384] | 0.716 [0.635 to 0.791]

11. Primary Outcome: Active Travel to School Based on Parental Report
Description: Active travel to school (ATS) refers to the behaviour of travelling to school by human-powered means as opposed to motorised transportation, for example by walking or cycling. This was based on parental ATS reports.
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: Reports of ATS from parent and from child at baseline (week 0) and weekly during the post-randomisation period (week 1-8); ATS trips=active trips to school. This data is from all trips reported by the parent whether child ATS reports are available for the same days or not; this differs from N trips in 'Agreement Between Parent and Child Reports'
Measure: Number; unit: % ATS trips
Units Other Than Participants: total N trips to school (parent-reported
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (total N trips to school (parent-reported) | 382 | 597
% ATS trips
  % ATS trips reported by parent at baseline | 59.0 | 69.4
  % ATS trips reported by parent at endline (week 8) | 58.6 | 82.1

12. Primary Outcome: Active Travel to School Based on Child Report
Description: Percentage of active trips to school based on child report. This data is from all the trips reported by children, whether parental reports exist for the same day or not. For that reason, this differs from the number of trips reported in 'Agreement Between Parent and Child Reports' because in that case, both parent and child reports were required for the same day.
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: Children in Year 5 (age 9-10); reports of ATS were collected from the parent and from the child at baseline (week 0) and weekly during the post-randomisation period (week 1 to 8); ATS trips=active trips to school. This data are only from child reports of ATS.
Measure: Number; unit: % ATS trips
Units Other Than Participants: N trips to school reported by child
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N trips to school reported by child) | 634 | 516
% ATS trips
  % ATS trips reported by child at baseline | 86.4 | 82.2
  % ATS trips reported by child at endline (week 8) | 94.0 | 86.3

13. Primary Outcome: Differences in MVPA During the Times Reported by the Parent, Based on Parental Report
Description: differences in minutes of moderate-to-vigorous physical activity (MVPA) between ATS and non-ATS trips during the times reported by the parent as pertaining to the journey to school, based on parental report (i.e. parent reported whether the trip was ATS or non-ATS)
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: Trips to school reported, irrespective of the school where they were reported. No comparisons between control and intervention school due to the low number of non-active trips. Number of Participants Analyzed in the "ATS Trips" Arm is the total N of participants whose parents reported ATS and provided data for MVPA. Likewise for "Non-ATS Trips".
Measure: Mean (Standard Deviation); unit: minutes of MVPA
Units Other Than Participants: trips to school
Groups:
- ATS Trips: active trips to school
- Non-ATS Trips: non-active trips to school (e.g. car trips)
Arm/Group | ATS Trips | Non-ATS Trips
Number analyzed (Participants) | 24 | 7
Number analyzed (trips to school) | 99 | 13
minutes of MVPA | 2.46 (2.83) | 0.76 (0.95)
Statistical Analysis 1: Comparison: ATS Trips vs Non-ATS Trips; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); U=390.5 Z=-2.3 p=0.02 The mean and SD values are provided for descriptive purposes only

14. Primary Outcome: Differences in MVPA During the Hour Before the Classes, Based on Parental Report
Description: differences in MVPA between ATS and non-ATS trips during the hour before the classes (7:56-8:55), based on parental report (i.e. parent reported whether trip was ATS or non-ATS)
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: This outcome refers to trips to school reported, irrespective of the school where they were reported. There are no comparisons between control and intervention school due to the low number of non-active trips.
Measure: Mean (Standard Deviation); unit: minutes of MVPA
Units Other Than Participants: trips to school
Arm/Group | ATS Trips | Non-ATS Trips
Number analyzed (Participants) | 24 | 8
Number analyzed (trips to school) | 104 | 19
minutes of MVPA | 4.99 (4.11) | 2.55 (1.69)
Statistical Analysis 1: Comparison: ATS Trips vs Non-ATS Trips; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney) — U=665.5 Z=-2.3 p=0.02 The mean and SD values are provided for descriptive purposes only

15. Primary Outcome: Differences in MVPA During the Times Reported by the Parent, Based on Child Report
Description: differences in minutes of MVPA between ATS and non-ATS trips during the times reported by the parent as pertaining to the journey to school, based on child report (i.e. child reported whether trip was ATS or non-ATS)
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: minutes of MVPA
Units Other Than Participants: trips to school
Arm/Group | ATS Trips | Non-ATS Trips
Number analyzed (Participants) | 27 | 8
Number analyzed (trips to school) | 128 | 15
minutes of MVPA | 2.40 (2.68) | 0.81 (0.87)
Statistical Analysis 1: Comparison: ATS Trips vs Non-ATS Trips; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney) — U=596.5 Z=-2.4 p=0.02 The mean and SD values are provided for descriptive purposes only

16. Primary Outcome: Differences in MVPA During the Hour Before the Classes, Based on Child Report
Description: differences in minutes of MVPA between ATS and non-ATS trips during the hour before the classes (7:56-8:55), based on child report (i.e. child reported whether trip was ATS or non-ATS)
Time Frame: 9 weeks (one week at baseline plus eight weeks after baseline)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: minutes of MVPA
Units Other Than Participants: trips to school
Arm/Group | ATS Trips | Non-ATS Trips
Number analyzed (Participants) | 28 | 10
Number analyzed (trips to school) | 146 | 20
minutes of MVPA | 4.99 (3.91) | 2.59 (1.60)
Statistical Analysis 1: Comparison: ATS Trips vs Non-ATS Trips; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney) — U=955.0 Z=-2.5 p=0.01 The mean and SD values are provided for descriptive purposes only

17. Primary Outcome: Parental ATS Reports by SMS
Description: Number of parental ATS reports by SMS.
  * In this case, for comparability with data from paper reports, one SMS reports refers to a week in which at least one SMS report was received from the parent.
  * Parental SMS reports were only possible in those weeks when the child was not wearing the accelerometer. Parents who had chosen to report ATS by SMS were requested to report by paper on the weeks when the child wore the accelerometer (once at baseline, and once at post-baseline), and could report ATS by SMS in all other weeks.
Time Frame: 8 weeks after baseline
Population: - 'One SMS report' refers to a week in which at least one SMS report of ATS was received from the parent throughout the study. The above 'number of units analyzed' refers to the total number of weeks, for all participants, in which parents could have reported ATS throughout the study.
Measure: Number; unit: N weeks with at least one SMS reply
Units Other Than Participants: N weeks with at least one SMS reply
Arm/Group | Intervention Group School | Control Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N weeks with at least one SMS reply) | 53 | 56
N weeks with at least one SMS reply | 51 | 56

18. Secondary Outcome: Number of Participants Who Met Physical Activity Guidelines
Description: Number of participants who met physical activity guidelines, i.e. at least 60 minutes of moderate-to-vigorous physical activity (MVPA) a day, measured by accelerometer (ActiGraph GT3X+); cut points of intensity by Evenson et al (2008) (sedentary <100 counts per minute (cpm); light >100cpm; moderate >=2296cpm; vigorous >=4012cmp), epoch 10 seconds. Valid wear was at least 6h/day on at least 3 days (weekdays or weekends).
  NOTE: the above criterion of 10h/day for at least 5 days was changed before the start of the fieldwork, although not on this website. We found studies which suggested that wearing the accelerometer 6h/day on at least three days, with or without weekend days, were sufficient to assess overall levels of physical activity. Consistent with these findings, this new minimum wear criterion was adopted in the present study.
Time Frame: 9 weeks
Population: 14 participants in the control school (2 dropouts after baseline) and 15 in the intervention school (0 dropouts). Participants wore the accelerometer twice in the study, for one week each time. N of valid recordings= N children who met the minimum wear target (6h/day on at least 3 days) overall; only valid recordings were used to assess overall PA
Measure: Number; unit: N children who met PA guidelines
Units Other Than Participants: N of valid recordings available overall
Arm/Group | Control Group School | Intervention Group School
Number analyzed (Participants) | 14 | 15
Number analyzed (N of valid recordings available overall) | 19 | 27
N children who met PA guidelines | 3 | 3

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Control Group School | Intervention Group School
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
* Few resources available to recruit schools and families
* Small sample size
* Small number of non-ATS trips with MVPA data
* The same person delivered the intervention, collected and analysed the data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No